CLINICAL TRIAL: NCT00296010
Title: Phase III Trial Evaluating the Role of Adjuvant Pegylated Liposomal Doxorubicin (PLD, Caelyx, Doxil) for Women (Age 66 Years or Older) With Endocrine Nonresponsive Breast Cancer Who Are Not Suitable for Being Offered a " Standard Chemotherapy Regimen"
Brief Title: Liposomal Doxorubicin Compared With Observation or Cyclophosphamide and Methotrexate in Treating Older Women Who Have Undergone Surgery for Breast Cancer
Acronym: CASA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Accrual rate was too low
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000463710; IBCSG-32-05 (Other: IBCSG); BIG-CASA (Other: Breast International Group); 2005-003434-18 (EudraCT Number); BIG-1-05 (Other: Breast International Group); EU-205112
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Methotrexate; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CASA-nil PLD (Experimental): Adjuvant pegylated liposomal doxorubicin (PLD) for 16 weeks
  Interventions: Drug: pegylated liposomal doxorubicin hydrochloride; Procedure: adjuvant therapy; Radiation: radiation therapy
- CASA-Nil (Active Comparator): No adjuvant therapy
  Interventions: Radiation: radiation therapy
- CASA-CM PLD (Experimental): Adjuvant pegylated liposomal doxorubicin (PLD) for 16 weeks
  Interventions: Drug: pegylated liposomal doxorubicin hydrochloride; Procedure: adjuvant therapy; Radiation: radiation therapy
- CASA-CM CM (Active Comparator): Low-dose, metronomic cyclophosphamide and methotrexate (CM) for 16 weeks
  Interventions: Drug: cyclophosphamide; Drug: methotrexate; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide — cyclophosphamide 50 mg/day orally continuously for 16 weeks
  Arms: CASA-CM CM
Drug: methotrexate — methotrexate 2.5 mg twice a day orally on days 1 and 4 of every week for 16 weeks
  Arms: CASA-CM CM
Drug: pegylated liposomal doxorubicin hydrochloride — Caelyx (R) (Doxil (R)) 20 mg/m2 iv x 8 doses (delivered every 2 weeks)
  Arms: CASA-CM PLD; CASA-nil PLD
Procedure: adjuvant therapy
  Arms: CASA-CM CM; CASA-CM PLD; CASA-nil PLD
Radiation: radiation therapy — Radiation therapy should be used according to institutional accepted guidelines. Radiation therapy to the conserved breast is recommended. Radiation therapy to the chest wall following mastectomy is optional (if given, it may also include nodal fields). Radiation therapy may be given either during operation or after all chemotherapy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate, cyclophosphamide, and liposomal doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether giving liposomal doxorubicin after surgery is more effective than observation or cyclophosphamide and methotrexate in treating breast cancer.

PURPOSE: This randomized phase III trial is studying liposomal doxorubicin to see how well it works compared with observation or cyclophosphamide and methotrexate in treating older women who have undergone surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the breast cancer-free interval in elderly women with resectable, hormone receptor-negative breast cancer treated with pegylated doxorubicin hydrochloride liposome (PDL) vs observation or PDL vs cyclophosphamide and methotrexate.

Secondary

* Compare the tolerability of these regimens in these patients.
* Compare the safety and toxic effects of these regimens in these patients.
* Compare the overall and progression-free survival of patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare the sites of failure in patients treated with these regimens.
* Compare the competing causes of death in patients treated with these regimens.
* Compare the rate of second non-breast malignancy in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are assigned, based on patient preference, to 1 of 2 treatment groups.

* Group 1: Patients are randomized to 1 of 2 arms (arms I and II).

  * Arm I: Patients receive pegylated doxorubicin hydrochloride liposome (PDL) IV over 1 hour on day 1. Treatment repeats every 2 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients undergo observation only.
* Group 2: Patients are randomized to 1 of 2 treatment arms (arms III and IV).

  * Arm III: Patients receive PDL as in arm I.
  * Arm IV: Patients receive oral cyclophosphamide once daily on days 1-7 and oral methotrexate twice daily on days 1 and 4. Treatment repeats every week for 16 courses in the absence of disease progression or unacceptable toxicity.

All patients may undergo radiotherapy according to institutional standards either during surgery or after the completion of chemotherapy.

Quality of life is assessed at baseline and at 3, 6, and 12 months.

After completion of study treatment, patients are followed periodically for 1 year.

PROJECTED ACCRUAL: A total of 1,296 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Disease must be confined to the breast and axillary nodes without detected masses elsewhere
  * No history of prior ipsilateral or contralateral invasive breast cancer
* Resected disease

  * No more than 16 weeks since last surgery to remove the tumor
  * No known clinical residual locoregional disease
  * Margins must be negative for invasive breast cancer and ductal carcinoma in situ
* No locally advanced, inoperable breast cancer including any of the following:

  * Inflammatory breast cancer
  * Supraclavicular node involvement
  * Enlarged internal mammary nodes unless pathologically negative
* Synchronous bilateral invasive breast cancer (diagnosed in the past 2 months) allowed if all tumors are hormone receptor-negative
* Must not be a candidate for endocrine therapy or standard chemotherapy
* Hormone receptor-negative disease

PATIENT CHARACTERISTICS:

* Female
* Menopausal status: postmenopausal
* ECOG performance status 0-2
* Platelet count ≥ 100,000/mm^3
* Granulocyte count ≥ 1,500/mm^3
* WBC ≥ 3,000/mm^3
* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin normal
* Creatinine clearance ≥ 50 mL/min
* Creatinine < 1.35 mg/dL
* No significant malabsorption syndrome or disease affecting gastrointestinal tract function
* No myocardial infarction within the past 6 months
* No pulmonary embolism within the past 6 months
* No deep vein thrombosis within the past 6 months
* No New York Heart Association class III or IV heart disease
* LVEF ≥ 50% by echocardiography, radionucleotide ventriculography, or MUGA
* No evidence of acute ischemia by ECG
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or bladder, or ipsilateral or contralateral breast carcinoma in situ
* No active, uncontrolled infection
* No active hepatitis B or C virus infection
* No other chronic infection
* Patients must not have any of the following "geriatric syndromes":

  * Dementia
  * Delirium
  * Major depression (as diagnosed by a psychiatrist)
  * Recent falls
  * Spontaneous bone fractures
  * Neglect
  * Abuse
* No evidence of medically relevant conduction system abnormalities that would preclude study entry
* No other nonmalignant, uncontrolled systemic diseases, psychiatric illness, or addictive or cognitive disorder that would preclude study participation or compliance

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior raloxifene, tamoxifen citrate, or other selective estrogen receptor modulators (SERMs)
* No concurrent recombinant human epoetin alfa or pegfilgrastim
* No prior neoadjuvant or adjuvant therapy for breast cancer except radiotherapy
* Concurrent trastuzumab (Herceptin®) allowed
* No concurrent hormonal replacement therapy
* No other concurrent hormonal therapy (including estrogen, progesterone, androgens, tamoxifen citrate, SERMs, or aromatase inhibitors) except for the following:

  * Steroids for adrenal failure
  * Hormones for non-disease-related conditions (e.g., insulin for diabetes)
  * Intermittent dexamethasone as an antiemetic
* No other concurrent investigational agents
* No concurrent bisphosphonates, except for the treatment of osteoporosis
* For patients who received prior anthracyclines, the following criteria must be met:

  * Cumulative dose ≤ 240 mg/m² for conventional doxorubicin

    * ≤ 140 mg/m² in case of prior doxorubicin and left chest radiotherapy (LCRT)
  * Cumulative dose ≤ 400 mg/m² for epirubicin

    * ≤ 230 mg/m² in case of prior epirubicin and LCRT

Ages: 66 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Breast cancer free interval by physical examination, laboratory tests, and investigations every 2 weeks for 16 weeks during treatment, every 3-6 months for 5 years, then annually as indicated after completion of study treatment | 5 years after recruitment starts

SECONDARY OUTCOMES:
Adverse events assessed by CTCAE v3.0 every 2 weeks for 16 weeks during treatment, every 3-6 months for 5 years, then annually after completion of study treatment | 5 years after recruitment starts
Quality of life assessed by Casa QL form, Mini-Cog, and VES-13 at baseline and at 2, 6, and 12 months after completion of study treatment | 5 years after recruitment starts
Disease-free survival by physical examination, laboratory tests, and investigations every 2 weeks for 16 weeks during treatment, every 3-6 months for 5 years, then annually as indicated after completion of study treatment | 5 years after recruitment starts
Overall survival by physical examination, laboratory tests, and investigations every 2 weeks for 16 weeks during treatment, every 3-6 months for 5 years, then annually as indicated after completion of study treatment | 5 years after recruitment starts
Sites of failure by physical examination, laboratory tests, and investigations every 2 weeks for 16 weeks during treatment, every 3-6 months for 5 years, then annually as indicated after completion of study treatment | 5 years after recruitment starts
Second (non-breast) malignancy by physical examination, laboratory tests, and investigations every 2 weeks for 16 weeks during treatment, every 3-6 months for 5 years, then annually as indicated after completion of study treatment | 5 years after recruitment starts
Causes of death prior to breast cancer recurrence by physical examination, laboratory tests, and investigations every 2 wks for 16 wks during treatment, every 3-6 mo. for 5 yrs, then annually as indicated after completion of study treatment | 5 years after recruitment starts

CONTACTS AND LOCATIONS:
Overall Officials: Diana Crivellari, MD, Study Chair — Centro di Riferimento Oncologico, Aviano (Italy); Silvia Dellapasqua, MD, Study Chair — European Institute of Oncology, Milano (Italy); Anne Hamilton, MD, Study Chair — Royal Prince Alfred Hospital, Camperdown (Australia)
Locations (33):
- Australia (4):
  - Gosford Hospital, Gosford, New South Wales
  - Nepean Cancer Care Centre at Nepean Hospital, Kingswood, New South Wales
  - Royal Hobart Hospital, Hobart, Tasmania
  - Frankston Hospital, Frankston, Victoria
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - Centre Hospitalier Etterbeek Ixelles, Brussels
  - AZ Groeninge - Oncologisch Centrum, Kortrijk
  - U.Z. Gasthuisberg, Leuven
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
- National Institute of Oncology, Budapest, Hungary
- Italy (11):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale degli Infermi - ASL 12, Biella
  - Ospedale Civile Ramazzini, Carpi
  - Ospedale Civile S. Croce, Fano
  - European Institute of Oncology, Milan
  - Ospedale Civile Rimini, Rimini
  - Ospedale Sant' Eugenio, Rome
  - Centro Sociale Oncologico, Treste
  - Policlinico Universitario Udine, Udine
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Auckland City Hospital, Auckland, New Zealand
- Institutul Oncologic - Universitatea de Medicina, Cluj-Napoca, Romania
- Institute of Oncology - Ljubljana, Ljubljana, Slovenia
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Skaraborgs Hospital, Skövde
- Switzerland (7):
  - Kantonspital Aarau, Aarau
  - Inselspital Bern, Bern
  - Oncocare Sonnenhof-Klinik Engeriedspital, Bern
  - Kantonsspital Graubuenden, Chur
  - Ospedale Beata Vergine, Mendrisio
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun